CLINICAL TRIAL: NCT04175171
Title: A Randomized, Double-blind, Parallel-group, Comparative Phase I Study to Evaluate the Safety and Pharmacokinetics of Single Intravenous (IV) Administration of GB221 Versus Herceptin® (Trastuzumab)
Brief Title: Clinical Trial of Comparative Study of GB221 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GB221-001
Record Dates: First submitted 2019-11-12; First posted 2019-11-22 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB221 (Experimental): Coprelotamab Injection, 8mg/kg, single dose
  Interventions: Drug: Coprelotamab Injection
- Herceptin (Active Comparator): Trastuzumab Injection, 8mg/kg, single dose
  Interventions: Drug: Trastuzumab Injection

INTERVENTIONS:
Drug: Coprelotamab Injection — The single intravenous infusion of 8mg/kg Coprelotamab shall be administered within 90 minutes through infusion pump.
  Other Names: GB221
  Arms: GB221
Drug: Trastuzumab Injection — The single intravenous infusion of 8mg/kgTrastuzumab shall be administered within 90 minutes through infusion pump.
  Other Names: Herceptin
  Arms: Herceptin

SUMMARY:
The primary objective is to assess the safety of a single dose of GB221 compared to Herceptin® when administered as a single IV injection at a dose of 8 mg/kg. The secondary objective of the study is to assess the pharmacokinetics of GB221 compared to Herceptin®.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, subjects must meet the following criteria

1. Males aged 18 to 45 years.
2. Healthy as judged by medical examination and medical history, and clinical chemistry and hematology screening.
3. Body weight within the normal range for height (BMI between 19.0 and 29.0, inclusive) up to a maximum of 90 kg.
4. Normal or non-clinically significant ECG.
5. Normotensive (systolic: 90 - 140; diastolic: 50 - 90 mm Hg, inclusive) and heart rate (40 -100 bpm, inclusive).
6. Willingness to give written and informed consent prior to any studyrelated procedures being conducted

Exclusion Criteria:

Subjects will be ineligible for the study if any of the following criteria apply:

1. Receipt of any investigational agent or drug within 4 weeks of entry to the study.
2. Use of any medicine - prescription, over-the-counter or herbal - in the 7 days prior to the treatment day and until 12 weeks after the treatment day.
3. Donation of blood (or loss of blood) greater than 400 ml within 3 months of the study.
4. Clinically significant drug allergy or sensitivity to any medication.
5. A history of chronic or recurrent infections.
6. A recent history of surgery.
7. History or presence of malignancy (with the exception of successfully treated basal cell carcinoma).
8. Inability to communicate or cooperate with the Principal Investigator because of English language difficulties or poor mental development.
9. A history (within the last 5 years) or evidence of alcohol or drug abuse (excepting tobacco use less than 10 cigarettes per day).
10. A positive urine test for drugs of abuse or alcohol either at screening or on the day of admittance for drug administration.
11. Vaccination of any type within the previous month.
12. A history of major psychiatric illness (such as bipolar disorder, schizophrenia or persistent major depression). Previous minor depression/adjustment disorder is acceptable if currently asymptomatic.
13. Consumption of more than 3 standard drinks per day, and not able to abstain from alcohol totally within 24 hours of dose administration.
14. Presence of current infection with tuberculosis, Hepatitis B, Hepatitis C or HIV.
15. History of asthma or other chronic respiratory disease in the past 5 years.
16. History of neurological or neuromuscular disease.
17. History of hypertension or cardiovascular disease, including congestive heart failure and cardiomyopathy or a clinically significant echocardiogram finding at the screening visit.
18. History of bladder or urethral disease.
19. Smoking cigarettes > 10 per day.
20. Any other condition which in the view of the Principal Investigator is likely to interfere with the study or put the subject at risk.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2012-01-08 (Actual); Study Completion 2012-03-08 (Actual)

PRIMARY OUTCOMES:
physical examination | Up to 84 days
  physical examination
adverse event | Up to 84 days
  adverse event
blood pressure | Up to 84 days
  blood pressure
heart rate | Up to 84 days
  heart rate
respiration rate | Up to 84 days
  respiration rate
oxygen saturation | Up to 84 days
  oxygen saturation
temperature | Up to 84 days
  temperature

SECONDARY OUTCOMES:
C max | Up to 84 days
  C max
t max | Up to 84 days
  t max
AUC | Up to 84 days
  AUC
CL | Up to 84 days
  CL
t ½ | Up to 84 days
  t ½
V | Up to 84 days
  V

CONTACTS AND LOCATIONS:
Overall Officials: Andrewn Redfer, PhD; MBBS, Principal Investigator — Linear Clinical Research Limited
Locations (1):
- Linear Clinical Research Limited, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No